CLINICAL TRIAL: NCT03815214
Title: Take Off Pounds After Stroke Trial (TOPS)
Acronym: TOPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Jennifer Dearborn-Tomazos, Assistant Professor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018P000770
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Stroke; Obesity; Overweight; Hemiparesis
MeSH Terms: conditions — Stroke; Obesity; Overweight; Paresis | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor is blinded to study group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet Intervention (Experimental): The diet intervention is a partial meal replacement program using the commercially available OPTAVIA® Optimal Weight 4&2&1 Plan™. In the OPTAVIA program, subjects are asked to eat 6 times each day, once every 2 to 3 hours.
  Interventions: Behavioral: Partial meal replacement program
- Enhanced Standard Care (Placebo Comparator): The control group will receive instruction on a healthy diet as defined by the United States Department of Agriculture.
  Interventions: Behavioral: Dietary Counseling

INTERVENTIONS:
Behavioral: Partial meal replacement program — Four meals consist of meal replacements made by OPTAVIA, such as shakes, soups, bars, biscuits, hot drinks, and puddings. Meal replacements will be provided to subjects without charge. For two other daily meals, subjects or their caregivers will be taught how to prepare meals consisting of 5-7 ounces (cooked) of a low-fat protein, 3 servings of non-starchy vegetables, and up to 2 servings of healthy fats.
  Arms: Diet Intervention
Behavioral: Dietary Counseling — Participants will receive one 45-minute counseling session on a healthy diet
  Arms: Enhanced Standard Care

SUMMARY:
The Take Off Pounds after Stroke (TOPS) trial is a Prospective Randomized Open-Label Blinded Endpoint (PROBE) study that will test a 12-week high protein, calorie restricted, partial meal replacement program, compared to enhanced standard care, for efficacy in achieving clinically significant weight loss without impairment of physical function patients with elevated body mass index (BMI) following a recent ischemic stroke.

DETAILED DESCRIPTION:
The TOPS trial is designed as a PROBE study to test the feasibility, safety, and efficacy of a 12-week high protein, calorie restricted, partial meal replacement program, compared to enhanced standard care, in achieving clinically significant weight loss without impairment of physical function when initiated within 90 days following ischemic stroke in patients with BMI 27-to-49.9 kg/m2.

Participants will be randomized in a 1-1 ratio to the partial meal replacement program (diet intervention) or enhanced standard care (control) with randomization stratified by recruitment center (BIDMC, Yale) and baseline diet consistency status (Modified Consistency Diet vs Regular Consistency Diet). Baseline diet consistency status was selected as a stratification factor because it is expected that patients with difficulty swallowing (dysphagia) after stroke that results in need for modifications to food/liquids will have a different weight loss trajectory than patients who are able to safely consume a regular diet. The follow-up duration will be 12 weeks for all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke within 90 days of randomization
2. Age >=18
3. BMI 27-49.9 mg/kg2
4. Able to meet all nutritional and fluid needs by oral intake.
5. Ready to undergo behavioral change
6. Able and willing to provide written informed consent
7. Maximum weight <=350 lbs

Exclusion Criteria:

1. Medical contraindication to weight loss or diet, including the following: renal disease requiring dialysis, taking lithium, or end stage liver or renal disease considered incompatible with diet intervention by patient's personal healthcare provider or the study PI
2. Enrollment in a conflicting clinical trial (defined as a trial with an intervention known to affect weight or with an exclusion for participation in another trial)
3. Pregnancy or desire to become pregnant, or currently breastfeeding
4. High-risk of malnutrition using a standard screen
5. Trajectory of recent weight loss (i.e., loss of at least 12 lbs in the 3 months preceding screening)
6. Allergy to soy based food products
7. Require thickening of liquids due to dysphagia
8. Inability to communicate with study team
9. Inability to speak English
10. Irreversible medical conditions likely to affect short-term survival (predicted survival of less than one year)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving at least a 5% weight loss | 12 weeks
  Proportion of subjects achieving at least a 5% weight loss from baseline to 12 weeks in the intervention group compared to the control group

OTHER OUTCOMES:
Change in blood pressure | 12 weeks
  Change in blood pressure from baseline to 12 weeks
Change in Waist Circumference | 12 weeks
  Change in waist circumference from baseline to 12 weeks
Change in Body Mass Index | 12 weeks
  Change in Body Mass Index from baseline to 12 weeks
Change in modified Rankin scale | 12 weeks
  Change in modified Rankin scale from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
The findings from this study will be presented at scientific meetings and published in scientific journals without revealing the identity of the subjects. The investigators plan to acknowledge the study subjects for their participation. The overall results of the study will be shared with the participants, accompanied by a thank you note, upon publication of the final results.

REFERENCES:
- [Result] Dearborn Tomazos J, Viscoli C, Amin H, Lovelett LJ, Rivera J, Gull A, Kernan WN. Partial Meal Replacement for Weight Loss after Stroke: Results of a Pilot Clinical Trial. Cerebrovasc Dis. 2024;53(1):54-61. doi: 10.1159/000530996. Epub 2023 May 15. PMID 37231793